CLINICAL TRIAL: NCT07239037
Title: Comparison Between TMJ Arthrocentesis Using the Dental Implant Motor Irrigation Pump and the Conventional Technique in Treatment of Internal Derangement
Brief Title: MJ Arthrocentesis Using the Dental Implant Motor Irrigation Pump and the Conventional Technique in Treatment of Internal Derangement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0911-05/2024
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: TMJ Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- implant motor irrigation I (Experimental)
  Interventions: Other: Motor irrigation with 80% power
- implant motor irrigation II (Experimental)
  Interventions: Other: Motor irrigation with 40% power
- Conventional arthrocentesis (Active Comparator)
  Interventions: Other: conventional TMJ arthrocentesis

INTERVENTIONS:
Other: Motor irrigation with 80% power — ten patients with TMJ internal derangement with reduction using dental implant motor irrigation pump in power 80%
  Arms: implant motor irrigation I
Other: Motor irrigation with 40% power — ten patients with TMJ internal derangement with reduction using dental implant motor irrigation pump in power 40%
  Arms: implant motor irrigation II
Other: conventional TMJ arthrocentesis — ten patients with TMJ internal derangement using conventional technique
  Arms: Conventional arthrocentesis

SUMMARY:
Background: Millions of individuals worldwide suffer from temporomandibular joint (TMJ) disorders and are characterized by pain and joint dysfunction. TMJ internal derangement (ID) is the most frequent type of temporomandibular disorders (TMDs). TMJ arthrocentesis represents a form of minimally invasive surgical treatment in patients suffering from internal derangement of the TMJ Aim of the study: To clinically compare between the effect of TMJ arthrocentesis under high hydraulic pressure by dental implant motor and the conventional method in treatment of TMJ internal derangement regarding pain and mandibular movements.

ELIGIBILITY:
Inclusion Criteria:

* TMJ internal derangement with reduction.
* Both genders.

Exclusion Criteria:

* Patients with overlying infection or cellulitis
* Relevant systemic disease
* Previous TMJ surgery.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Change in pain scores | 1 week, 4 weeks, 3 months
  a 10 point visual analogue scale (VAS)*. (0-1=none, 2-4=mild, 5-7=moderate, 8-10=severe) .
Change in mouth opening | baseline, 1 week, 4 weeks, 3 months
  The patient's maximum mouth opening (MMO) value will be measured by taking the average of three consecutive measurements of the distance between the maxilla and mandible mid-central incisive teeth with the Endo ruler after the patients were asked to open

SECONDARY OUTCOMES:
post operative edema | 1 week
  Scales:
  * None (no swelling)
  * Mild (intra oral swelling confined to surgical field)
  * Moderate (extra oral swelling in the surgical zone)
  * Severe (extra oral swelling spreading beyond the surgical zone)
change in mandibular movements | baseline, 1 week, 3 months
  Patient's TMJ Lateral, protrusive and side to side movements will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt